CLINICAL TRIAL: NCT05293340
Title: Avocado Voucher Impact on Health Outcomes in Hispanic/Latino Adults With or At-risk of Type 2 Diabetes
Brief Title: Continuous Glucose Monitoring and Hass Avocado Trial ("CHAT")
Acronym: CHAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per discretion of Sponsor.
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Hass Avocado Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C2021-0068
Record Dates: First submitted 2021-12-22; First posted 2022-03-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Dietary Habits; Diabetes Mellitus, Type 2
Keywords: Glycemic control; Minority Health; Plants, Edible; Food prescriptions; Food security; Time in Range
MeSH Terms: conditions — Feeding Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study will consist of two groups into which participants will be randomly assigned 1:1. One (active) group will receive vouchers for free avocados. The other (control) group will not receive avocado vouchers (to control for the impact of seasonal changes on diet that are outside the influence of the trial).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hispanic/Latino adults with or at risk of T2D- Active Group (Experimental): Eligible participants receive vouchers for free avocados.
  Interventions: Dietary Supplement: Avocado Vouchers
- Hispanic/Latino adults with or at risk of T2D- Control Group (No Intervention): Eligible participants will not receive vouchers for free avocados.

INTERVENTIONS:
Dietary Supplement: Avocado Vouchers — Food as Medicine to demonstrate clinically meaningful benefits for underserved communities. Avocados are fruits with fats, fiber, micronutrients, and bioactive phytochemicals.
  Arms: Hispanic/Latino adults with or at risk of T2D- Active Group

SUMMARY:
Hispanic/Latino adults in the United States (U.S.) bear a disproportionate burden of type 2 diabetes (T2D). Dietary changes, facilitated by increased access and adherence to healthy foods, are necessary. In this study, continuous glucose monitoring (CGM) will be used to quantify changes in glycemic control in Hispanic/Latino (predominantly of Mexican origin) adults with or at-risk of T2D before and after receiving free avocados for 12 weeks. Beyond CGM-measured glycemic control, wearable activity and sleep monitors, physical exams, laboratory analyses, and questionnaires/logs will be used to track the impact of free avocado vouchers. The findings are anticipated to help clinicians provide new information to support positive behavior change to reduce the risk of T2D or progression from pre-diabetes to T2D and make it easier for patients to access healthier food, potentially leading to improved health.

DETAILED DESCRIPTION:
In this study, continuous glucose monitoring (CGM) will be used to quantify changes in glycemic control in Hispanic/Latino adults with and at-risk of T2D before and after receiving free avocado vouchers. The impact of using CGM to determine the effect of improving access to avocados on glycemic profiles and food related-behaviors for Hispanic/Latino adults with or at risk of T2D is not known at present. To address this need, increased avocado consumption will be combined with CGM to assess post-prandial glucose responses. This is based on evidence showing that one half of a Hass avocado at lunch is associated with increased satisfaction and reduced desire to eat over the subsequent 3-5 hours in overweight or obese adults.

For CGM, there is a lack of prospective data on the relationship between derived metrics and complications for adults with non-insulin treated T2D or at-risk of T2D, but glucose profiles from non-diabetic subjects suggest very tight glycemic control, with only brief postprandial excursions >140 mg/dL. Cross-sectional data suggests more time spent between 140 and 180 mg/dl comparing predominantly Mexican American adults at risk of T2D to adults with pre-T2D and to adults with diagnosed T2D. Further, in a study examining the thresholds for CGM at which vascular disease can be detected, Lu and colleagues reported time in ranges above 140 mg/dL was associated with abnormal values for retinopathy and carotid intima-medial thickness, a measure of macrovascular disease risk. Hence, the focus in this study will be time in range between 140 and 180 mg/dl between 6 am and 12 am (waking hours).

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at enrollment.
2. Self-reported Hispanic/Latino heritage.
3. Self-reported diagnosis of T2D or self-reported as at risk for developing T2D using the American Diabetes Association diabetes risk assessment tool [25].

Exclusion Criteria:

1. Use of insulin
2. Pregnancy
3. Any active clinically significant disease or disorder which in the investigator's opinion could interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Time in range (TIR) between 140 and 180 mg/dL [TIR (140-180)]- Change from Prior to Intervention, to Final Two Weeks of Intervention | Prior to Intervention (Week 0), and During Final 2 Weeks of Intervention (Week 13 or 14)
  TIR (140 -180 mg/dL) between 6 am and 12 am (waking hours).

SECONDARY OUTCOMES:
Waist Circumference- Change from Enrollment Visit to Study Conclusion Visit | At Enrollment Visit and at 14 weeks from Enrollment Visit
  Changes in waist circumference
Blood Pressure- Diastolic and Systolic- Change from Enrollment Visit to Study Conclusion Visit | At Enrollment visit and at 14 weeks from Enrollment Visit
  Changes in blood pressure
HbA1c- Change from Enrollment Visit to Study Conclusion Visit | At Enrollment Visit and at 14 weeks from Enrollment Visit
  Changes in HbA1c
Insulin resistance- Change from Enrollment Visit to Study Conclusion Visit | At Enrollment visit and at 14 weeks from enrollment visit
  Changes in Insulin Resistance
Lipids- Change from Enrollment Visit to Study Conclusion Visit | At enrollment visit and at 14 weeks from enrollment visit
  Changes in lipids
Prescribed medicines for T2D and/or hypertension- Change from Enrollment Visit to Study Conclusion Visit | At enrollment visit and at 14 weeks from enrollment visit
  Changes in prescribed medicines for T2D and/or hypertension
Self-reported sleep, mood, and pain via 100 mm Likert scale questionnaire- Change from Enrollment, and to Final Visit | At enrollment visit, and at 14 weeks from enrollment visit
  Changes in self-reported sleep, mood, and pain (Best to Worst)
Self-reported Food security via United States Dept. of Agriculture U.S. Household Food Security Survey Module: Six-Item Short Form - Change from Enrollment, and at Final Visit | At enrollment visit, and at 14 weeks from enrollment visit
  Changes in Food Security
Depression via the Depression, Anxiety and Stress Scale (DASS-21) | At enrollment visit, and at 14 weeks from enrollment visit
  Change in depression score (0-42), with higher scores indicating higher levels of depression
Anxiety via the Depression, Anxiety and Stress Scale (DASS-21) | At enrollment visit, and at 14 weeks from enrollment visit
  Change in anxiety score (0-42), with higher scores indicating higher levels of anxiety
Stress via the Depression, Anxiety and Stress Scale (DASS-21) | At enrollment visit, and at 14 weeks from enrollment visit
  Change in stress score (0-42), with higher scores indicating higher levels of stress
Change in Eating Self-Efficacy Scale (ESES) score | Prior to intervention (Week 0), and during final 2 weeks of intervention (Week 13 or 14)
  Change in Eating Self-Efficacy Scale (ESES) mean score (25-175), with higher scores indicating lower eating self-efficacy.
Change in Self-Report Habit Index (SRHI) score | Prior to intervention (Week 0), and during final 2 weeks of intervention (Week 13 or 14)
  Change in Self-Report Habit Index (SRHI) mean score (1-7), with higher scores indicating stronger habits.
Change in Self-Regulation of Eating Questionnaire (SREBQ) score | Prior to intervention (Week 0), and during final 2 weeks of intervention (Week 13 or 14)
  Change in Self-Regulation of Eating Behaviour Questionnaire (SREBQ) mean score (1-5), with higher scores indicating better self-regulation of eating behavior.
Physical Activity- Daily step count, Changes from first to final Fitbit application | First Fitbit application (pre-intervention) to second Fitbit application (in final 14 days of intervention)
  Physical Activity- Daily step count averaged over ≤14 days, Change from first Fitbit application (pre-intervention) to second Fitbit application (in final 14 days of intervention).
Sleep Duration | First Fitbit application (pre-intervention) to second Fitbit application (in final 14 days of intervention)
  Change in Sleep Duration (in minutes) averaged over ≤14 days
Secondary Continuous Glucose Monitoring Endpoints- Time in Range (TIR) 140-180 mg/dl, Waking Hours | first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
  Change in TIR between 140 and 180 mg/dL [TIR (140-180)] between 6 am and 12 am (waking hours), averaged over ≤14 days from first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
Secondary Continuous Glucose Monitoring Endpoints- Average Glucose | first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
  Change in Average Glucose averaged over ≤14 days from first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
Secondary Continuous Glucose Monitoring Endpoints- Time in Range (TIR) 70-180 mg/dL | first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
  Change in TIR 70-180 mg/dL averaged over ≤14 days from first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
Secondary Continuous Glucose Monitoring Endpoints- Time >180 mg/dL | first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
  Change in time >180 mg/dL averaged over ≤14 days from first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
Secondary Continuous Glucose Monitoring Endpoints- Time <70 mg/dL | first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
  Change in time <70 mg/dL averaged over ≤14 days from first CGM application (pre-intervention) to second CGM application (in final 14 days of intervention).
Adherence to the intervention | 12-week intervention monitoring period running weeks 2-14
  Adherence to the intervention as measured via the daily avocado consumption log (DACL)
Acceptability of the intervention | 12-week intervention monitoring period running weeks 2-14
  Acceptability of the intervention as measured by the weekly avocado acceptability questionnaire (WAAQ)
Regression analysis between avocado adherence measured as an average number of avocados consumed as reported via the daily avocado consumption log (DACL) and personality traits assessed via the Mini International Personality Item Tool. | Average over 12 weeks
  Each participant will fill out the Mini International Personality Item Tool (Mini-IPIP) at the start of the study. It comprises 20 items and assesses the five personality factors (Extraversion, Agreeableness, Conscientiousness, Neuroticism, and Imagination). Scoring includes computing the mean score for each factor with a value ranging from 1 to 5 (very inaccurate to very accurate). Avocado adherence measured as the mean of the number of avocados consumed as reported via the daily avocado consumption log (DACL) will be computed. A regression analysis will be performed between the mean of the number of avocados consumed as the response variable and the five personality factors scores as the predictor variables. The coefficients of the regression analysis will be studied to evaluate if personality traits can predict avocado adherence.
Regression analysis between the average number of avocados consumed as reported via the daily avocado consumption log (DACL) and motives underlying the selection of food assessed by the Food Choice Questionnaire (FCQ) | Average over 12 weeks
  Each participant will fill out the Food Choice Questionnaire at the start of the study. It comprises 36 items and assesses the importance of 9 types of motives underlying food selection (Health, Mood, Convenience, Sensory Appeal, Natural Content, Price, Weight Control, Familiarity and Ethical Concern). Scoring includes computing the mean score for each type of motive ranging from 1-4 with higher values indicating higher importance. Avocado adherence measured as the mean of the number of avocados consumed as reported via the daily avocado consumption log (DACL) will be computed. A regression analysis will be performed between the mean of the number of avocados consumed as the response variable and the scores of the 9 types of motives underlying food selection as the predictor variables. The coefficients of the regression analysis will be studied to evaluate if food choice motives can predict avocado adherence.
Regression analysis between average composite acceptability score on the weekly Avocado Acceptability Questionnaire and Personality traits assessed via the Mini International Personality Item Tool. | Average over 12 weeks
  Each participant will fill out the Mini International Personality Item Tool at the start of the study. It comprises 20 items and assesses the five personality factors (Extraversion, Agreeableness, Conscientiousness, Neuroticism, and Imagination). Scoring includes computing the mean score for each factor with a value ranging from 1 to 5 (very inaccurate to very accurate). The mean of the composite acceptability score on the weekly Avocado Acceptability Questionnaire (average taken over 12 weeks) will be computed. A regression analysis will be performed between the mean of the composite acceptability score as the response variable and the five personality factors scores as the predictor variables. The coefficients of the regression analysis will be studied to evaluate if personality traits can predict acceptability score.
Regression analysis between average composite acceptability score on the weekly Avocado Acceptability Questionnaire and motives underlying the selection of food assessed by the Food Choice Questionnaire (FCQ) | Average over 12 weeks
  Each participant will fill out the Food Choice Questionnaire at the start of the study. It comprises 36 items and assesses the importance of 9 types of motives underlying food selection (Health, Mood, Convenience, Sensory Appeal, Natural Content, Price, Weight Control, Familiarity, and Ethical Concern). Scoring includes computing the mean score for each type of motive ranging from 1-4 with higher values indicating higher importance. The mean of the composite acceptability score on the weekly Avocado Acceptability Questionnaire (average taken over 12 weeks) will be computed. A regression analysis will be performed between the mean of the composite acceptability score as the response variable and the scores of the 9 types of motives underlying food selection as the predictor variables. The coefficients of the regression analysis will be studied to evaluate if food choice motives can predict acceptability score.

CONTACTS AND LOCATIONS:
Overall Officials: David Kerr, MBChB, Principal Investigator — Sansum Diabetes Research Institute
Locations (1):
- Sansum Diabetes Research Institute, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No